CLINICAL TRIAL: NCT03570229
Title: Pelvic Radiation Injuries After Cancer Treatment: Symptoms, Quality of Life and Experiences Before, Along and After Hyperbaric Oxygenation Treatment
Brief Title: Hyperbaric Oxygenation Treatment and Quality of Life
Status: Completed | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, May Aasebø Hauken, Prinsipal Investigator, University of Bergen
Other Study IDs: 01012018
Record Dates: First submitted 2018-05-02; First posted 2018-06-26 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Cancer
Keywords: Quality of life (QOL); Hyperbaric oxygen treatment (HBOT); Late radiation tissue injury (LRTI); Longitudinal; Mixed methods; Patient experiences
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Hyperbaric oxygen treatment — Participants in this study will receive hyperbaric oxygen treatment (HBOT) but the investigators do not assign this specific intervention to the study participants. Thus, the patients in this study will receive HBOT as part of routine medical care. Consequently, we regard this as an observational study because the patients will get HBOT independently of the study and they are NOT assigned prospectively to HBOT according to a protocol to evaluate the effects.
  HBOT for pelvic radiation injury typically involves a treatment pressure of 2.4 ATA (Atmospheres Absolute) breathing oxygen for 90 minutes. The treatment is delivered as series treatment, usually daily treatment up to 30 dives.

SUMMARY:
Osteoradionecrosis, dermal soft tissue necrosis, radiation cystitis, proctitis and sexual dysfunctions are well-known late-effects after radiation for cancer in the pelvic area, negatively affecting the survivors' quality of life (QOL) and psychosocial wellbeing. Increasing evidence and clinical practice support the use of hyperbaric oxygen treatment (HBOT) as an effective treatment in a variety of radiation injuries, but this is still a field with limited research and knowledge. Especially, there is a knowledge gap on how late radiation tissue injury (LRTI) influences cancer survivors' QOL and psychosocial health in a longitudinal perspective (before, along and after HBOT), as well as the patients' knowledge, expectation and experience from this treatment. This study aims to improve knowledge on these issues.

DETAILED DESCRIPTION:
Late effects following radiation of pelvic cancers:

Annually, more than 32000 Norwegians are diagnosed with cancer where approximately 70% will be alive 5 years after diagnosis. About 50% of all cancer patients receive radiation as part of their multimodal cancer treatment, and 50% of these will be long-term survivors. Irradiation therapy is an essential part of the curative treatment of pelvic malignancies, including rectal, uterine and cervical carcinoma. Although precautions and advances are taken, radiation may affect surrounding healthy tissue and lead to acute or chronic radiation injury. About 5-15% of the patients experience late radiation tissue injury (LRTI) that develops months or years after radiation, characterized by poor microcirculation with hypoxia, tissue damage and fibrosis. Consequently, frequent late-effects are related to radiation cystitis, proctitis and enteritis, soft tissue necrosis (skin and vagina) and fistulas with increased frequency, urgency and leakage of urine or faces, diarrhoea and pain. Although these late- effects obviously interfere significantly with the survivors' quality of life (QOL) and psychosocial health, research regarding these consequences is extremely limited.

Hyperbaric oxygen treatment (HBOT) for pelvic LRTI:

HBOT is a treatment modality where the patient is placed in a pressure chamber breathing 100% oxygen while exposed to elevated ambient pressure. HBOT for pelvic LRTI typically involves a treatment pressure of 2.4 ATA Atmospheres Absolute) while breathing oxygen once daily for about 90 minutes for 6 weeks (about 30 'dives' in total). HBOT for LRTI is based upon its ability to increase tissue oxygenation, stimulate neoangiogenesis and cellular regeneration and thereby induce revitalizing and healing of damaged tissue. Although HBOT is a time- consuming treatment, it is well accepted and tolerated by the patients, with few and usually harmless side effects.

Previous studies on the effect of HBOT to reduce pelvic LRTI have not yet yielded broadly accepted and conclusive results. The available studies indicate that HBOT has a positive effect on a variety of conditions, although some studies report no effect. A Cochrane review concludes that HBOT may improve outcomes in various kinds of cancer related radiation injuries (e.g. head and neck, proctitis, osteoradionecrosis), suggesting that other tissues also are likely to respond (e.g. bladder). However, these studies operate with very heterogeneous timepoints for follow-up, varying from right after HBOT is finished to several weeks, months or years after, which may have influenced the outcomes. However, we could not find any publication stating the course of symptomatic improvement for pelvic LRTI. This knowledge-gap is a challenge when informing patients and handling their expectations for this treatment.

QOL following HBOT:

Late-effects from cancer treatment, especially pelvic LRTI, may affect all parts of cancer survivors' life. Consequently, quality of life (QOL) is reckoned as an important outcome as it comprises physiological, psychological and social aspects of well-being. However, there is an evident research gap on how pelvic LRTI influences the patients' QOL, as well as how these outcomes develop in a longitudinal perspective. Two studies show QOL improvement in patients with chronic diabetic foot ulcers after 6 weeks. One study found significant QOL improvements from perioperative HBOT in the dimensions of pain, global health and dyspnoea in 66 patients with head and neck cancers. Another study of 101 radiation-injured patients (54% head and neck, 36 % intestine and 11% bladder) showed significant one-year improvements in the QOL dimensions of vitality and physical-, role- and social function. A significantly improved healing and increased bowel-specific QOL was found immediately after HBOT and at one-year follow-up in a randomized controlled study of 120 patients with radiation proctitis. In contrast, a systematic review state that no conclusion about HBOT's influence on QOL can be made.

In summing up, different outcomes of HBOT from pelvic radiation injured cancer survivors in a longitudinal perspective are highly requested as the existing research comprises small samples, has methodological limitations and yields scant results.

The study's goals and research questions:

This study embraces three main goals: The primary goal is to improve knowledge on how QOL is affected in survivors of pelvic cancer with LRTI, and how this may change due to HBOT. The second goal is to gain information on the patients' knowledge and expectations concerning HBOT and their experiences and satisfaction with the care along the HBOT process. The third goal is to improve knowledge on the longitudinal changes in LRTI symptoms and the patients' long-term QOL after finishing HBOT. Consequently, this study addresses the following research questions:

1. How do patients experience that the LRTI symptoms influence their everyday life?
2. What perceived information, knowledge and expectations concerning HBOT do patients express before HBOT?
3. What are the patients' self-reported LRTI burden,QOL and psychosocial health before HBOT?
4. How do LRTI symptoms change during and after the HBOT course?
5. How do QOL and psychosocial health change during the HBOT course?
6. What is the correlation between LRTI symptoms and QOL during and after the HBOT process?
7. How do patients experience the HBOT process?
8. How satisfied with care are patients along the HBOT process, and which factors do they describe as important for their satisfaction?
9. What are the patients' long-term QOL, psychosocial health and LRTI burden after HBOT?

Study design:

Based on the research questions, we will perform a mixed methods study with a prospective longitudinal embedded design. Mixed method is reckoned as the third research paradigm, and in this design quantitative data are collected longitudinal (> 3 time-points) and qualitative data are collected at two time points. This design is especially recommended where randomization is not suited or possible, and because it draws on the strengths and minimalizes the weaknesses of both quantitative and qualitative methods. Consequently, it may yield a more complete and nuanced picture of the topic, as validated questionnaires provide quantitative outcome data and in-depth interviews provide process data to explore and elaborate the quantitative results.

Recruitment and eligibility criteria: The study will recruit participants from patients that have been referred to HBOT and will undergo the treatment independently from the study. Participation in the study will neither influence whether patients are treated with HBOT, nor time or lengths or any other HBOT-related measure.

Data collection: see elsewhere

Analyses of data:

Quantitative analyses: Statistical tests will be two-tailed, with statistical significance defined as P< .05. Descriptive statistics, correlations, paired T-tests, multiple regression analyses and longitudinal analysis with linear mixed models (LMM) (or the equvalent non-Parametric tests dependent of the characteristics of the final data set) will be used for analysis of change. Effect sizes will be calculated by Cohen's d, while Z tests will be performed to analyze differences between the sample mean and the mean in the general populations.

Qualitative analysis: Systematic text condensation (STC) will be used to analyze qualitative data. This is a descriptive and exploratory method for thematic cross-case analysis of interviews. STC is a four-step analysis that includes 1) gaining a total impression; 2) identifying units of meaning; 3) abstracting the contents of individual units of meaning; 4) summarizing their importance.

Ethics:

The Regional Committee for Medical and Health Research Ethics in northern Norway has approved the project (2018/706). The study will be conducted in line with the Helsinki Declaration, providing the participants with oral and written information and written consent. As all participants will be treated with HBOT independent of inclusion in the study, we do not anticipate any negative outcomes for study-patients.

Project management, organization and cooperation:

This study is a cooperation between Center for Crisis Psychology (CCP), Faculty of Psychology, University of Bergen and Section for Hyperbaric Medicine (SHM), Department of Occupational Medicine (DOM), at Haukeland University Hospital in Bergen, Norway. A project group, chaired by CCP's research leader, May Hauken, will run the project. As HBOT represents a narrow field internationally, the study is connected to DOM's already existing international partners in the Nordic cooperation. Additionally, a multidisciplinary and international Advisory Board will be connected to the project. User involvement will be include throughout the study and include patients, representative from the Norwegian Gynecological Cancer Organization and health care professionals working with HBOT.

Progress plan and dissemination of results:

This is a 4 year project with a specific progress plan. Based on the research questions and collected data, we plan to publish at least 8 scientific papers in international peer-reviewed journals. Results will also be disseminated via lectures, popular scientific papers, national and international conferences. At the end of the project period, we will arrange a summing -up conference.

ELIGIBILITY:
Inclusion Criteria:

1. pelvic radiation injury after intended curative radiation therapy for pelvic cancer (prostate, gynecological, and urological and bowel cancers),
2. ≥ 6 months from finished radiation therapy
3. referred to the unit for hyperbaric oxgen treatment (HBOT)
4. aged ≥ 18 years.

Exclusion Criteria:

1. severe physical and/or mental co-morbidity representing a contraindication for HBOT
2. insufficient cognitive or language skills to answer study questionnaires and perform interviews.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit participants from all patients with pelvic radiation injury assigned to oxygen treatment (HBOT) at Section for Hyperbaric Medicine (SHM) at Haukeland University Hospital in Bergen, being the Norwegian National Center for planned HBOT.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life after HBO-therapy | Change from baseline (T1) to 30 weeks (T7, 6 months after end of HBO-therapy)
  Self reported quality of life scale, European Organization for Research and Treatment of Cancer (EORTC QLQ C30) scale, 30 questions, 4-point Likert scale 0-3 for 28 items, 0-6 for two items, total score 0-100 (100=highest level of functioning/ best score)

SECONDARY OUTCOMES:
Long-term change in Quality of life | Change from baseline (T1) to 58 weeks (T8, 1 year after end of HBO-therapy)
  Self reported quality of life scale, European Organization for Research and Treatment of Cancer (EORTC QLQ C30) scale, 30 questions, 4-point Likert scale 0-3 for 28 items, 0-6 for two items, total score 0-100 (100=highest level of functioning/ best score)
Change in Late radiation tissue injury symptoms after HBO-therapy | Change from baseline (T1) to 30 weeks (T7, 6 months after end of HBO-therapy)
  Expanded Prostate Cancer Index (EPIC) questionnaire, urinary (12 items) and bowel (14 items) subscores, 3- to 5-point Likert scale, sum-score 0-100 (0=worst symptoms)
Time to improvement in Late radiation tissue injury symptoms | Time from baseline (T1) to significant improvement (at least 0,5 SD) up to 30 weeks (T7) after end of HBO-therapy
  Expanded Prostate Cancer Index (EPIC) questionnaire, urinary (12 items) and bowel (14 items) subscores, 3- to 5-point Likert scale, sum-score 0-100 (0=worst symptoms), improvement defined as a higher score of at least 0,5 standard deviations based on the study population
Satisfaction With Care | T3 (after 6 weeks)
  Total score of EORTC in-PATSAT 32 (European Organization of Research and Treatment of Cancer, In-patient satisfaction With care), 32 questions, 5-point Likert scale, total score 0-100, higher score = more satisfied with care

CONTACTS AND LOCATIONS:
Overall Officials: May Aa Hauken, Professor, Study Chair — University of Bergen
Locations (1):
- University of Bergen/Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Yes
We plan to make IPD available to other researchers on NSD (Norwegian Scientific Data).
Supporting Information: Study Protocol
Time Frame: After the study has finished, earliest in December 2022
Access Criteria: On request

REFERENCES:
- [Background] Niezgoda JA, Serena TE, Carter MJ. Outcomes of Radiation Injuries Using Hyperbaric Oxygen Therapy: An Observational Cohort Study. Adv Skin Wound Care. 2016 Jan;29(1):12-19. doi: 10.1097/01.ASW.0000473679.29537.c0. PMID 26650092
- [Background] Viswanathan AN, Lee LJ, Eswara JR, Horowitz NS, Konstantinopoulos PA, Mirabeau-Beale KL, Rose BS, von Keudell AG, Wo JY. Complications of pelvic radiation in patients treated for gynecologic malignancies. Cancer. 2014 Dec 15;120(24):3870-83. doi: 10.1002/cncr.28849. Epub 2014 Jul 23. PMID 25056522
- [Background] Do NL, Nagle D, Poylin VY. Radiation proctitis: current strategies in management. Gastroenterol Res Pract. 2011;2011:917941. doi: 10.1155/2011/917941. Epub 2011 Nov 17. PMID 22144997
- [Background] Plafki C, Carl UM, Glag M, Hartmann KA. The treatment of late radiation effects with hyperbaric oxygenation (HBO). Strahlenther Onkol. 1998 Nov;174 Suppl 3:66-8. PMID 9830461
- [Background] Gorenstein S, Katz A, Regan K, Hangan D. A retrospective case series looking at the effectiveness of hyperbaric oxygen in treating radiation cystitis. Journal of Clinical Oncology. 2015;33(7_suppl):127-127.
- [Background] Cancer Registry of Norway. Cancer in Norway 2015 - Cancer incidence, mortality, survival and prevalence in Norway. Oslo: Cancer Registry of Norway; 2016.
- [Background] Weir G. Hyperbaric oxygen therapy for complications of radiotherapy. Wound Healing South Africa. 2009;2(2):60-62.
- [Background] Jaeger K, Juttner B, Franko W. [Hyperbaric oxygen therapy--options and limitations]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2002 Jan;37(1):38-42. doi: 10.1055/s-2002-20080. No abstract available. German. PMID 11845381
- [Background] Macdonald HM. Hyperbaric oxygenation in the patient with malignancy: friend or foe? Diving and Hyperbaric Medicine. 2007;37(3):133-138.
- [Background] Camporesi EM. Side effects of hyperbaric oxygen therapy. Undersea Hyperb Med. 2014 May-Jun;41(3):253-7. PMID 24984321
- [Background] Ennis RD. Hyperbaric oxygen for the treatment of radiation cystitis and proctitis. Curr Urol Rep. 2002 Jun;3(3):229-31. doi: 10.1007/s11934-002-0069-5. PMID 12084193
- [Background] Spiegelberg L, Djasim UM, van Neck HW, Wolvius EB, van der Wal KG. Hyperbaric oxygen therapy in the management of radiation-induced injury in the head and neck region: a review of the literature. J Oral Maxillofac Surg. 2010 Aug;68(8):1732-9. doi: 10.1016/j.joms.2010.02.040. Epub 2010 May 20. PMID 20493616
- [Background] Bennett MH, Feldmeier J, Hampson NB, Smee R, Milross C. Hyperbaric oxygen therapy for late radiation tissue injury. Cochrane Database Syst Rev. 2016 Apr 28;4(4):CD005005. doi: 10.1002/14651858.CD005005.pub4. PMID 27123955
- [Background] Safra T, Gutman G, Fishlev G, Soyfer V, Gall N, Lessing JB, Almog R, Matcievsky D, Grisaru D. Improved quality of life with hyperbaric oxygen therapy in patients with persistent pelvic radiation-induced toxicity. Clin Oncol (R Coll Radiol). 2008 May;20(4):284-7. doi: 10.1016/j.clon.2007.12.005. Epub 2008 Jan 28. PMID 18222656
- [Background] Oscarsson N, Arnell P, Lodding P, Ricksten SE, Seeman-Lodding H. Hyperbaric oxygen treatment in radiation-induced cystitis and proctitis: a prospective cohort study on patient-perceived quality of recovery. Int J Radiat Oncol Biol Phys. 2013 Nov 15;87(4):670-5. doi: 10.1016/j.ijrobp.2013.07.039. Epub 2013 Sep 11. PMID 24035333
- [Background] van Ophoven A, Rossbach G, Pajonk F, Hertle L. Safety and efficacy of hyperbaric oxygen therapy for the treatment of interstitial cystitis: a randomized, sham controlled, double-blind trial. J Urol. 2006 Oct;176(4 Pt 1):1442-6. doi: 10.1016/j.juro.2006.06.065. PMID 16952654
- [Background] Chong V, Rice M. The effectiveness of hyperbaric oxygen therapy (HBOT) in radiation-induced haemorrhagic cystitis. N Z Med J. 2016 Dec 2;129(1446):79-83. PMID 27906922
- [Background] Ferreira C, Reis F, Correia T, et al. Hyperbaric oxygen for long-term complications of radiation cystitis. Journal of Radiotherapy in Practice. 2014;14(1):18-26.
- [Background] Craighead P, Shea-Budgell MA, Nation J, Esmail R, Evans AW, Parliament M, Oliver TK, Hagen NA. Hyperbaric oxygen therapy for late radiation tissue injury in gynecologic malignancies. Curr Oncol. 2011 Oct;18(5):220-7. doi: 10.3747/co.v18i5.767. PMID 21980249
- [Background] Glover M, Smerdon GR, Andreyev HJ, Benton BE, Bothma P, Firth O, Gothard L, Harrison J, Ignatescu M, Laden G, Martin S, Maynard L, McCann D, Penny CEL, Phillips S, Sharp G, Yarnold J. Hyperbaric oxygen for patients with chronic bowel dysfunction after pelvic radiotherapy (HOT2): a randomised, double-blind, sham-controlled phase 3 trial. Lancet Oncol. 2016 Feb;17(2):224-233. doi: 10.1016/S1470-2045(15)00461-1. Epub 2015 Dec 17. PMID 26703894
- [Background] Carr JA, Higginson IJ, Robinson PG. Quality of life. London: BMJ Books; 2003.
- [Background] Crosby RD, Kolotkin RL, Williams GR. Defining clinically meaningful change in health-related quality of life. J Clin Epidemiol. 2003 May;56(5):395-407. doi: 10.1016/s0895-4356(03)00044-1. PMID 12812812
- [Background] Londahl M, Landin-Olsson M, Katzman P. Hyperbaric oxygen therapy improves health-related quality of life in patients with diabetes and chronic foot ulcer. Diabet Med. 2011 Feb;28(2):186-90. doi: 10.1111/j.1464-5491.2010.03185.x. PMID 21219427
- [Background] Li G, Hopkins RB, Levine MAH, Jin X, Bowen JM, Thabane L, Goeree R, Fedorko L, O'Reilly DJ. Relationship between hyperbaric oxygen therapy and quality of life in participants with chronic diabetic foot ulcers: data from a randomized controlled trial. Acta Diabetol. 2017 Sep;54(9):823-831. doi: 10.1007/s00592-017-1012-z. Epub 2017 Jun 12. PMID 28603808
- [Background] Harding SA, Hodder SC, Courtney DJ, Bryson PJ. Impact of perioperative hyperbaric oxygen therapy on the quality of life of maxillofacial patients who undergo surgery in irradiated fields. Int J Oral Maxillofac Surg. 2008 Jul;37(7):617-24. doi: 10.1016/j.ijom.2008.04.004. Epub 2008 May 23. PMID 18501562
- [Background] Clarke RE, Tenorio LM, Hussey JR, Toklu AS, Cone DL, Hinojosa JG, Desai SP, Dominguez Parra L, Rodrigues SD, Long RJ, Walker MB. Hyperbaric oxygen treatment of chronic refractory radiation proctitis: a randomized and controlled double-blind crossover trial with long-term follow-up. Int J Radiat Oncol Biol Phys. 2008 Sep 1;72(1):134-143. doi: 10.1016/j.ijrobp.2007.12.048. Epub 2008 Mar 14. PMID 18342453
- [Background] Lauvrak V, Fronsdal KB, Ormstad SS, Vaagbo G, Fure B. Effectiveness of Hyperbaric Oxygen Therapy in Patients with Late Radiation Tissue Injury or Diabetic Foot Ulcer [Internet]. Oslo, Norway: Knowledge Centre for the Health Services at The Norwegian Institute of Public Health (NIPH); 2015 Mar. Report from Norwegian Knowledge Centre for the Health Services (NOKC) No. 4-2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK390572/ PMID 28510406
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Creswell JW, Clark VL. Designing and conducting mixed method research. London: SAGE Publications, Inc.; 2011.
- [Result] Velure GK, Muller B, Hauken MA. Symptom burden, psychological distress, and health-related quality of life in cancer survivors with pelvic late radiation tissue injuries. Support Care Cancer. 2022 Mar;30(3):2477-2486. doi: 10.1007/s00520-021-06684-x. Epub 2021 Nov 15. PMID 34779920
- [Result] Hauken MA, Velure GK, Muller B, Sekse RJT. Sexual Health and Quality of Life in Cancer Survivors With Pelvic Radiation Injuries. Cancer Nurs. 2024 Sep-Oct 01;47(5):E298-E307. doi: 10.1097/NCC.0000000000001259. Epub 2023 Jul 14. PMID 37449715
- [Result] Velure GK, Muller B, Hauken MA. Symptom burden and health-related quality of life six months after hyperbaric oxygen therapy in cancer survivors with pelvic radiation injuries. Support Care Cancer. 2022 Jul;30(7):5703-5711. doi: 10.1007/s00520-022-06994-8. Epub 2022 Mar 23. PMID 35320424
- [Result] Velure GK, Müller B, Aa. Hauken M. Experiences of patients with pelvic radiation injuries after cancer treatment undergoing hyperbaric oxygen therapy: A phenomenological-hermeneutical study. Nordic Journal of Nursing Research. 2021;41(3):131-9.